CLINICAL TRIAL: NCT01282853
Title: The Influence of Biopsy Number and Site on the Sensitivity of Rapid Urease Test for Diagnosis of H. Pylori Infection in Patients With Bleeding Gastroduodenal Ulcer
Brief Title: Rapid Urease Test for Diagnosis of H. Pylori Infection in Patients With Peptic Ulcer Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzong-Hsi Lee, M.D., Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FEMH-99-C-029
Record Dates: First submitted 2011-01-23; First posted 2011-01-25 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2011-01

CONDITIONS: Peptic Ulcer; Hemorrhage
Keywords: peptic ulcer; hemorrhage; rapid urease test; urea breath test
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Active Comparator): one biopsy specimen taken from gastric antrum was put into RUT kit
  Interventions: Procedure: endoscopic biopsy
- A4 (Experimental): 4 biopsy specimens taken from gastric antrum were put into RUT kit
  Interventions: Procedure: endoscopic biopsy
- B1 (Experimental): one biopsy specimen taken from gastric body was put into RUT kit
  Interventions: Procedure: endoscopic biopsy

INTERVENTIONS:
Procedure: endoscopic biopsy — endoscopic biopsy for rapid urease test
  Other Names: HelicotecUT plus for rapid urease test
  Arms: A1
Procedure: endoscopic biopsy — endoscopic biopsy for rapid urease test
  Other Names: HelicotecUT plus for rapid urease test
  Arms: A4
Procedure: endoscopic biopsy — endoscopic biopsy for rapid urease test
  Other Names: HelicotecUT plus for rapid urease test
  Arms: B1

SUMMARY:
Rapid urease test (RUT) is the most commonly used biopsy-based method to diagnose Helicobacter pylori (Hp) infection because of its simple, rapid and accurate characters. However, its sensitivity was reported to decrease during ulcer bleeding recently. So it is an important issue to avoid a false negative test in these patients. Siddique et al reported that the sensitivity of RUT could be increased when the biopsy number increased from 1 to 4. Other studies demonstrated that additional biopsy from gastric body would increased the sensitivity of RUT in patients with ulcer bleeding. Therefore, we design this study to see if increased number of biopsy or different location of biopsy could increase sensitivity of RUT in patients with gastroduodenal ulcer bleeding.

After receiving explanation and giving consent, these patients with gastric or duodenal ulcer bleeding diagnosed after endoscopic examination will be enrolled. Those who are unstable, have received antibiotic or continuous proton pump inhibitor treatment within 4 weeks, or are contraindicated for endoscopic biopsy will be excluded. We will take 1 piece, 4 pieces of biopsy samples from prepyloric antrum and 1 piece from gastric body with standard biopsy forceps from the patients after they agree for RUT test. Then, we put these samples into 3 separate RUT kits respectively. We use 13C-UBT as gold standard for diagnosis of Hp infection. It is scheduled: (1) if the condition of this patient is not suitable for breath test just after endoscopic examination, 13C-UBT will be performed within 2 days,(2) otherwise, it will be performed 1 hour after examination. We plan to enroll 100 patients for this study. We will apply McNamer's test to examine the difference of RUT sensitivity of different biopsy number. For the RUT sensitivity from different locations, we use kappa statistic method to analyze their consistency.

DETAILED DESCRIPTION:
as brief summary

ELIGIBILITY:
Inclusion Criteria:

* gastroduodenal ulcer with bleeding, documented by endoscopic examination

Exclusion Criteria:

* 1. receiving continuous proton pump inhibitor treatment, antibiotics within 4 weeks 2. not suitable for endoscopic biopsy 3. hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the sensitivity of rapid urease test for H. pylori | within 2 days
  the sensitivity of rapid urease test for H. pylori using 13C-UBT as gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Tzong-Hsi Lee, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan, Taiwan